CLINICAL TRIAL: NCT04151277
Title: PRIMUS 001: An Adaptive Phase II Study of FOLFOX-A (FOLFOX and Nab-paclitaxel) Versus AG (Nab-paclitaxel and Gemcitabine) in Patients With Metastatic Pancreatic Cancer, With Integrated Biomarker Evaluation
Brief Title: PRIMUS 001: A Study Looking at Two Different Chemotherapy Regimens in Patients With Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Judith Dixon-Hughes (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); University of Glasgow (Other)
Responsible Party: Sponsor-Investigator, Judith Dixon-Hughes, Project Manager, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIMUS0012016
Record Dates: First submitted 2019-10-25; First posted 2019-11-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Neoplasms Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Albumin-Bound Paclitaxel; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to each of the treatments 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOX-A (Experimental): * nab-paclitaxel: 150mg/m2 IV over 30 minutes, day 1 (administered first)
  * Oxaliplatin: 85mg/m2, IV over 2 hours, day 1
  * Folinic acid: 350 mg flat dose, IV over 2 hours, day 1
  * 5-FU infusion:1200mg/m2/day, as a continuous IV infusion over 2 days, day 1 and day 2 (for a total dose of 2400mg/m2 over 46 hours (or 48 hours as per standard practice))
  Interventions: Drug: FOLFOX-A; Drug: G-CSF
- Abraxane and Gemcitabine (Active Comparator): * nab-paclitaxel: 125 mg/m2 IV over 30 minutes, day 1, 8, and 15 (administered first)
  * Gemcitabine 1000 mg/m2 IV over 30 minutes on days 1, 8, and 15 (immediately following nab-paclitaxel)
  Interventions: Drug: Gemcitabe and Abraxane

INTERVENTIONS:
Drug: FOLFOX-A — Patients will recieve nab-paclitaxel, oxaliplatin, Folinic Acid and 5-FU in a 14 day cycle
  Arms: FOLFOX-A
Drug: Gemcitabe and Abraxane — Patients will receive gemcitabine and nab-paclitaxel 3 weeks out of 4
  Arms: Abraxane and Gemcitabine
Drug: G-CSF — Patients in the FOLFOX-A arm will also receive daily G-CSF as primary prophylaxis for all cycles. This will be given as per local site policy for 14 day chemotherapy regimens
  Arms: FOLFOX-A

SUMMARY:
This study is comparing two combinations of chemotherapy treatments in patients with metastatic pancreatic cancer. Half the participants will receive FOLFOX-A and the other half will receive AG. Treatment will continue until progression or patient/clinican decision or intolerable toxicity.

DETAILED DESCRIPTION:
PRIMUS 001 is a multicentre, randomised, open label, two arm, phase II interventional trial with pre-clinical and translational work including in-depth molecular profiling and biomarker discovery/development. The primary objective is to look at the efficacy of FOLFOX-A compared to AG in all comers and in a biomarker positive group using progression free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been enrolled in the Precision-Panc Master Protocol
2. Patient has provided signed information consent for the PRIMUS 001 study
3. Age ≥ 16 years
4. Histologically-confirmed pancreatic ductal adenocarcinoma and its varients
5. Measurable metastatic disease according to RECIST V1.1
6. Eastern Cooperative Oncology Group (ECOG) 0-1 with life expectation of no less than 12 weeks
7. Patients must have received no previous chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with a fluoropyrimidine and/or gemcitabine administered in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no ongoing toxicities are present
8. Adequate liver/bone marrow function as defined by:

   1. Neutrophils (ANC) ≥ 1.5 x 109/l
   2. Platelets ≥ 100 x 109/l
   3. Haemoglobin ≥ 9.0 g/dL
   4. White Blood Cells (WBC) ≥ 3 x 109/l
   5. Total bilirubin ≤ 1.5 x institutional ULN unless bilirubin rise is due to Gilbert's syndrome
   6. Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN ( <5 ULN in the presence of liver metastases)
   7. Estimated creatinine clearance ≥ 60 mL/min (as calculated by Cockcroft and Gault or Wright formula or measured by EDTA clearance) 9. Negative serum or urine Human Chorionic Gonadotropin (HCG) test for females with child bearing potential. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential 10. Woman of child bearing potential, and men with female partners of child bearing potential, must agree to use adequate contraceptive measures (see s section 8.1.8.1) for the duration of the study and for up to 6 months after the completion of study treatment. 11. Compliant, and can be followed up regularly

The following additional inclusion criteria is ONLY required if recommended by the independent Data Monitoring Committee after interim review of study data (sites will have been informed by the Cancer Research UK (CRUK) Clinical Trials Unit (CTU) if this is the case) 12. Patient must be biomarker positive as fed back after central Precision-Panc diagnostic testing

Exclusion Criteria:

1. Prior treatment with nab-paclitaxel or oxaliplatin
2. Prior chemotherapy for metastatic pancreatic cancer
3. Known hypersensitivity for any component of any study drug
4. Active infection including Herpes Zoster and chickenpox
5. Current neuropathy ≥ grade 2
6. Uncontrolled brain metastasis
7. Uncontrolled congestive heart failure (CHF), or history of myocardial ischemia (MI), unstable angina, stroke, or transient ischemia within previous 6 months
8. Uncontrolled serious contraindicated medical condition or illness
9. Known or suspected dihydropyrimidine dehydrogenase (DPD) deficiency
10. Pregnant or breastfeeding
11. History of physical or psychiatric disorder that would prevent informed consent and compliance with protocol
12. Administration of any investigational drug within 28 days or 5 half-lives, whichever is longer, of receiving the first dose of trial treatment
13. Any systemic anti-cancer therapy or major surgery within 28 days of randomisation
14. Any minor surgery or radiotherapy within 7 days of randomisation
15. Any psychological, familial, sociological or geographical consideration potentially hampering compliance with the trial protocol and follow up schedule
16. Any patients receiving treatment with brivudin, sorivudin and analogues
17. History of another malignancy in the last 5 years (other than treated squamous/basal cell skin cancer, treated early-stage cervical cancer or treated/biochemically-stable organ-confined prostate cancer)
18. Any patient with severe diarrhoea (defined as ≥grade 3 diarrhoea despite maximum supportive measures and exclusion of underlying infection)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | At time of progression (estimated to be between 5 and 7.5 months)
  Progression free survival as measured froim the date of randomisation to progression or death (from any cause)

SECONDARY OUTCOMES:
Ojective Response Rate | Measured every 8 weeks by CT scan (most patients will received 3-4 CT scans over 24-32 weeks))
  Based on RECIST version 1.1
Overall Survival | From date of randomisation until date of death from any cause. Most patients with metastatic pancreatic cancer will die within 6-9 months from diagnosis
  Survival will be measured from the date of randomisation and include all caused of death
Safety and Tolerability of FOLFOX-A treatment | At every chemotherapy visit (every 2 weeks) - and at end of treatment visit (within 30 days of completing chemotherapy). Chemotherapy will continue until progression (estimated at between 5-7.5 months)
  Using NCI-CTCAE version 4.03
Safety and Tolerability of AG treatment | At every chemotherapy visit (3 weeks out of every 4) - and at end of treatment visit (within 30 days of completing chemotherapy). Chemotherapy will continue until progression (estimated at between 5-7.5 months)
  Using NCI-CTCAE version 4.03
Quality of Life (EORTC QLQ-C30) | Every 8 weeks while on treatment, at end of treatment visit, which will take place within 30 days of completing treatment, and at follow-up visits (6, 9, 12, 18, 24, 36, 48 and 60 months post randomisation).
  patients will complete the EORTC QLQ-C30 questionnaire at clinic
Peripheral Neuropathy | Every 4 weeks while on treatment, at end of treatment visit and at follow-up visits (6, 9, 12, 18, 24, 36, 48 and 60 months post randomisation).
  Measured by GOG-NTX4
Health Economics as defined to hospital resource use i.e how many nights the patient has spent in hospital and how may times they have attended hospital since the last time they were seen | At each study visit. Patient will be followed up for up to 5 years post randomistation (6, 9, 12, 18, 24, 36, 48 and 60 months post randomisation).
  Resource use will be assessed during the course of the study
Biomarker Discovery and Development | Ongoing during study. Recruitment will take 46 months and patients will be followed-up for up to 5 years post randomisation
  This will be ongoing as part of the study. This will use trial material but will be extrinsic to the trials outcomes. The biomarker will be specificed and locked down before the first interim analysis that is biomarker dependent
Quality of Life (EORTC QLQ-PAN26) | Every 8 weeks while on treatment, at end of treatment visit, which will take place within 30 days of completing treatment, and at follow-up visits (6, 9, 12, 18, 24, 36, 48 and 60 months post randomisation).
  patients will complete the EORTC QLQ-PAN26 questionnaire at clinic
Quality of Life (EQ-5D-5L) | Every 8 weeks while on treatment, at end of treatment visit, which will take place within 30 days of completing treatment, and at follow-up visits (6, 9, 12, 18, 24, 36, 48 and 60 months post randomisation).
  patients will complete the EQ-5D-5L questionnaire at clinic

CONTACTS AND LOCATIONS:
Overall Officials: Janet Graham, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (30):
- United Kingdom (30):
  - Aberdeen Royal Infirmary, Aberdeen
  - Northern Ireland Cancer Centre, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Castle Hill Hospital, Cottingham
  - Ninewells Hospital, Dundee
  - Western General, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Huddersfield Royal Infirmary, Huddersfield
  - Raigmore Hospital, Inverness
  - St James's University Hospital, Leeds
  - The Clatterbridge Cancer Centre, Liverpool
  - Guy's Hospital, London
  - Imperial College Healthcare Trust, London
  - Royal Free London Hospital, London
  - Royal Marsden Hospital, London
  - St Bart's Hospital, London
  - St George's Hospital, London
  - University College London Hospital, London
  - The Christie, Manchester, Manchester
  - Milton Keynes General Hospital, Milton Keynes
  - Freeman Hospital, Newcastle
  - Nottingham University Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Poole Hospital, Poole
  - Weston Park, Sheffield
  - University of Southampton Hospital, Southampton
  - Singleton Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, once the study report has been written and published, the anonymised clinical data will be available via request to Trial Management Group
Supporting Information: Study Protocol, CSR
Time Frame: After publication of study
Access Criteria: On Request to Trial Management Group